CLINICAL TRIAL: NCT05639036
Title: Image-guided External Ventricular Drain Placement Trial: a Prospective Randomized-controlled Trial Pilot
Brief Title: Image Guided EVD Placement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited resources available. Study unable to begin.
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 15534
Record Dates: First submitted 2022-11-09; First posted 2022-12-06 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-03

CONDITIONS: External Ventricular Drain (EVD); Image Guidance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-Free Hand External Ventricular Drain Placement (Active Comparator): This group will receive an external ventricular drain placed using the standard free-hand technique
  Interventions: Procedure: Free Hand External Ventricular Drain Placement
- Intervention - Image Guided External Ventricular Drain Placement Using the NAV3 System (Experimental): This group will receive an external ventricular drain placed using the assistance of the Stryker NAV3 image guidance system
  Interventions: Device: Image Guided External Ventricular Drain Placement Using the NAV3 System

INTERVENTIONS:
Device: Image Guided External Ventricular Drain Placement Using the NAV3 System — Nav3 image guidance system used to assist with external ventricular drain placement
  Arms: Intervention - Image Guided External Ventricular Drain Placement Using the NAV3 System
Procedure: Free Hand External Ventricular Drain Placement — External ventricular drain will be placed with the standard free-hand technique
  Arms: Control-Free Hand External Ventricular Drain Placement

SUMMARY:
To determine if use of the Stryker Nav3 image guidance system offers superior results in external ventricular drain (EVD) placement compared to the standard free-hand technique.

DETAILED DESCRIPTION:
An external ventricular drain (EVD) is a small tube that is placed into a space in the brain called a ventricle. This is done to drain fluid in the brain that sometimes builds up as a result of surgery or a traumatic brain injury/accident. This is one of most commonly performed procedures in Neurosurgery and is done bedside, not in the operating room. Typically, surgeons will use the "free-hand" technique to place these drains which involves relying on a CT scan, which shows the structures inside of the brain, and their knowledge of the anatomy of the brain and where the EVD should be placed. Image-guidance systems exist which create real time imaging of the patients brain and can act like a GPS to help guide the placement of the EVD in the correct spot. This trial is planned to determine if using the image guidance system does offer improved accuracy in EVD placement, lowering the number of attempts required and therefore the amount of time spent placing the EVD and risk of complications and infections. A pilot study will be done first, using a convenience sample at the Hamilton General Hospital to determine the feasibility of running a larger scale trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring EVD placement
* patients who can safely and reasonably be randomized to either study arm
* patients with available pre-procedural head CT
* written/verbal consent obtained

Exclusion Criteria:

* patients with very small ventricles/distorted ventricular anatomy from traumatic brain injury (ie it is not reasonable to randomize the patient)
* scenarios where the EVD must be inserted immediately and there is not time to obtain consent
* scenarios where bedside image guidance system (NAV3) is unavailable
* subjects medically or neurologically unstable to obtain pre-EVD CT scan
* EVD revisions on ipsilateral side during same admission

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Study Feasibility | 8 months
  Patient recruitment rate (patients/month), eligibility of patients (included/excluded), unexpected events (rate of occurrence)

SECONDARY OUTCOMES:
Accuracy of external ventricular drain (EVD) placement | 8 months
  Use of Kakarla grading system. This system uses a scale of 1 to 3, with 1 being optimal/satisfactory EVD placement, 2 being suboptimal EVD placement with the tip being placed in non-eloquent tissue, and 3 being suboptimal EVD placement with the tip being placed in eloquent tissue.
Number of attempts | 8 months
  Number of attempts required to satisfactorily place the EVD
Complications | 8 months
  Occurrence of any complications or infections will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kesava Reddy, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Patient data will be de-identified and the data will be analyzed as a whole before becoming available to other researchers.
  De-identified IPD may be shared with other researchers if necessary based on occurrence of adverse events occurrence, circumstantial findings, etc.

REFERENCES:
- [Background] Kakarla UK, Kim LJ, Chang SW, Theodore N, Spetzler RF. Safety and accuracy of bedside external ventricular drain placement. Neurosurgery. 2008 Jul;63(1 Suppl 1):ONS162-6; discussion ONS166-7. doi: 10.1227/01.neu.0000335031.23521.d0. PMID 18728595
- [Background] Aljoghaiman M, Bergen B, Takroni R, Wang B, Eangles P, Farrokhyar F, Sharma S. Image-Guided versus Freehand Ventricular Drain Insertion: Systematic Review and Meta-analysis. World Neurosurg. 2022 Apr;160:85-93.e5. doi: 10.1016/j.wneu.2022.01.036. Epub 2022 Jan 13. PMID 35033689